CLINICAL TRIAL: NCT05639140
Title: A Registered Observational Cohort Study on Color Discrimination Deficit Associated With Neurodegenerative Disorders.
Brief Title: A Registered Cohort Study on Color Discrimination Deficit Associated With Neurodegenerative Disorders.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort-Visual
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Neurodegenerative Disorders
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Color discrimination deficit
  Interventions: Other: Data collection
- Without Color discrimination deficit
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Neuropsychological assessment, FM-1OO, brain MRI, electroencephalogram and biomarker datas will be collected

SUMMARY:
Color discrimination deficit is a common manifestation of Alzheimer's disease (AD). However, the pathophysiology of this dysfunction remains poorly understood. The aim of the present study was to evaluate color discrimination using the Farnsworth-Munsell 100 hue test in patients with AD and mild cognitive impairment (MCI), compared with age-matched control subjects. As a secondary aim, we evaluated whether the outcomes of these visual tests were associated with cognitive.

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent extensive clinical examination including thorough neurological and somatic examination by a specialized neurologist or geriatrician and extensive neuropsychological examination by a trained psychologist. AD was diagnosed according to the NINCDS-ADRDA criteria.

Exclusion Criteria:

* We excluded individuals with noncompensated somatic illnesses, a history of a psychiatric disorder, color blindness, ophthalmological pathology, severe cranial trauma, focal neurological signs or magnetic resonance imaging examinations suggestive of cerebrovascular disturbances.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients include who suffer from Neurodegenerative Disorders whether Color discrimination deficit or not.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
MoCA scores | Baseline
  The Montreal Cognitive Assessment (MoCA)

SECONDARY OUTCOMES:
ACE-III scores | Baseline
  Addenbrooke's Cognitive Examination (ACE) score

OTHER OUTCOMES:
TES | Baseline
  The total error score

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No